CLINICAL TRIAL: NCT02886442
Title: A Pilot Evaluation of Adhesives and How They Are Impacted by Output
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_03
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-08

CONDITIONS: Ileostomy-stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 3 (Experimental): This is a sub-study testing how the adhesion of two adhesives is influenced by exposure to real output.
  There are two kinds of visits:
  Visit 1:
  Two adhesive strips (standard adhesive strip) are applied on the peristomal skin; one strip is exposed to real output (contained in a sleeve) and the other strip is not.
  Visit 2:
  Two adhesive strips (new adhesive strip) are applied on the peristomal skin; one strip is exposed to real output (contained in a sleeve) and the other strip is not.
  Visit 2:
  Interventions: Other: Standard adhesive strip; Other: New adhesive strip

INTERVENTIONS:
Other: Standard adhesive strip — This is a standard adhesive strip (hydrocolloid)
Other: New adhesive strip — This is a newly developed adhesive strip

SUMMARY:
This study investigates the impact of real output on the adhesion of two adhesives.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had an ileostomy for more than one year
4. Have intact skin on the area used in the evaluation
5. Has an ileostomy with a diameter up to (≤) 35 mm
6. Have a peristomal area accessible for application of patches/adhesive strips (assessed by investigating scientist) -

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Having dermatological problems in the peristomal- or abdominal area (assessed by investigating scientist)
5. Participating in other interventional clinical investigations or have previously participated in this evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Peel force | 12 hours
  The peel force was measured when the adhesive was removed

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Nielsen, MSc, Principal Investigator — Senior R&D scientist
Locations (1):
- Coloplast A/S, Humlebæk, Denmark